CLINICAL TRIAL: NCT02996253
Title: Endoscopic Assisted Transfer of Flexor Hallucis Longus Tendon for Chronic Achilles Tendon Rupture. A Prospective Multi Center Cohort Study
Brief Title: Endoscopic Transfer of Flexor Hallucis Longus Tendon for Chronic Achilles Tendon Rupture
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Central Hospital, Fredrikstad (Unknown)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, MD, PhD, Oslo University Hospital
Other Study IDs: 2015/16389
Record Dates: First submitted 2016-12-07; First posted 2016-12-19 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: FHL transfer — endoscopic transfer og flexor hallucis longus

SUMMARY:
The transfer of Flexor Hallucis Longus (FHL) in the management of chronic Achilles tendon ruptures has demonstrated good functional outcome, but an extensive surgical field at a vulnerable location may lead to increased risk for soft tissue problems. The arthroscopic FHL transfer may reduce the risk for soft tissue problems. Functional outcome parameters are investigated, wound/soft tissue complications registered.

DETAILED DESCRIPTION:
The transfer of FHL in the management of chronic Achilles tendon ruptures has demonstrated good functional outcome with American Orthopaedic Foot ane Ankle Society (AOFAS) hindfoot scores at 80-89. The extensive surgical field by either a two-incision approach or a single longitudinal posterior approach to the Achilles tendon may lead to an increased risk for soft tissue problems, both infections and wound healing problems. The endoscopic FHL transfer may reduce the risk for soft tissue problems while retaining a good functional outcome. Several functional outcome measures and scores are evaluated a year after surgery.

Prospective study for evaluation of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Achilles Tendon Rupture

Exclusion Criteria:

* Pregnancy
* BMI<18.5 or >39.9
* Insufficient Norwegian Language proficiency lack of communication skills local skin conditions at site for planned surgery

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With chronic Achilles Tendon Rupture
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-12; Primary Completion 2022-02 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The Victorian Institute of Sports Assessment- Achilles Questionnaire (VISA-A) outcome score | one year after FHL transfer

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain (VAS pain) score | 3, 6 and 12 months after FHL transfer
  patient reported outcome
patient reported function score (PRFS) | 6, 12 months
  patient reported Activity related disability
Magnetic resonance imagine (MRI) | one year post surgery
  FHL hypertrophy
functional test battery | 12 months
  jump- and strength tests
local wound conditions | within 12 weeks
  wound infection
AOFAS hindfoot | 3,6,12 months
VISA-A | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth E Husebye, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No